CLINICAL TRIAL: NCT02849080
Title: Efficacy and Safety of Oral Semaglutide Using a Flexible Dose Adjustment Based on Clinical Evaluation Versus Sitagliptin in Subjects With Type 2 Diabetes Mellitus
Acronym: PIONEER 7
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4257; 2015-005593-38 (EudraCT Number); U1111-1177-5103 (Other: WHO)
Record Dates: First submitted 2016-07-21; First posted 2016-07-29 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide flexible dosing (3, 7 or 14 mg) (Experimental)
  Interventions: Drug: semaglutide
- Sitagliptin 100 mg (Active Comparator)
  Interventions: Drug: sitagliptin

INTERVENTIONS:
Drug: semaglutide — Oral administration once-daily.
  Arms: Semaglutide flexible dosing (3, 7 or 14 mg)
Drug: sitagliptin — Oral administration once-daily.
  Arms: Sitagliptin 100 mg

SUMMARY:
This trial is globally conducted. The aim of this trial is to investigate Efficacy and Safety of Oral Semaglutide Using a Flexible Dose Adjustment Based on Clinical Evaluation versus Sitagliptin in Subjects with Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

Main phase (the inclusion criteria for the main phase are not reassessed for the extension phase):

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Male or female, age above or equal to 18 years at the time of signing informed consent. For Korea only: Male or female, age above or equal to 19 years at the time of signing informed consent
* Diagnosed with type 2 diabetes mellitus for at least 90 days prior to day of screening
* HbA1c (glycosylated haemoglobin) 7.5-9.5% (58-80 mmol/mol) (both inclusive)
* Treatment target of HbA1c below 7.0% (53 mmol/mol), as judged by the investigator
* Stable daily dose(s) of 1-2 of the following anti-diabetic drugs within 90 days prior to the day of screening:
* Metformin (equal or above 1500 mg or maximum tolerated dose as documented in the subject medical record)
* Sulfonylureas (equal or above half of the maximum approved dose according to local label or maximum tolerated dose as documented in subject medical record)
* Sodium glucose co-transporter 2 inhibitors
* Thiazolidinediones (equal or above half of the maximum approved dose according to local label or maximum tolerated dose as documented in subject medical record)

Extension phase:

* Informed consent for the extension phase obtained before any trial-related activities for the extension phase.
* On randomised treatment with or without rescue medication at week 52.

Exclusion Criteria:

Main phase (the exclusion criteria for the main phase are not reassessed for the extension phase):

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (adequate contraceptive measure as required by local regulation or practice). For certain specific countries: Additional specific requirements apply
* Any disorder, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol
* Family or personal history of Multiple Endocrine Neoplasia Type 2 or Medullary Thyroid Carcinoma
* History of pancreatitis (acute or chronic)
* History of major surgical procedures involving the stomach potentially affecting absorption of trial product (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery)
* Any of the following: myocardial infarction, stroke or hospitalisation for unstable angina or transient ischaemic attack within the past 180 days prior to the day of screening and randomisation
* Subjects presently classified as being in New York Heart Association Class IV
* Planned coronary, carotid or peripheral artery revascularisation known on the day of screening
* Subjects with alanine aminotransferase above 2.5 x upper normal limit
* Renal impairment defined as Estimated Glomerular Filtration rate 60 mL/min/1.73 m^2 as per Chronic Kidney Disease Epidemiology Collaboration formula
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria in a period of 90 days before the day of screening. An exception is short-term insulin treatment for acute illness for a total of below or equal to 14 days
* Proliferative retinopathy or maculopathy requiring acute treatment. Verified by fundus photography or dilated fundoscopy performed within 90 days prior to randomisation
* History or presence of malignant neoplasms within the last 5 years (except basal and squamous cell skin cancer and carcinoma in situ)
* History of diabetic ketoacidosis

Extension phase: There are no new exclusion criteria for the extension phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2016-09-20 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2019-03-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (73):
- United States (36):
  - Novo Nordisk Investigational Site, Glendale, Arizona
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Lancaster, California
  - Novo Nordisk Investigational Site, West Hills, California
  - Novo Nordisk Investigational Site, Boynton Beach, Florida
  - Novo Nordisk Investigational Site, Lake Worth, Florida
  - Novo Nordisk Investigational Site, Miami Lakes, Florida
  - Novo Nordisk Investigational Site, Port Orange, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Blackfoot, Idaho
  - Novo Nordisk Investigational Site, Evanston, Illinois
  - Novo Nordisk Investigational Site, Greenfield, Indiana
  - Novo Nordisk Investigational Site, Muncie, Indiana
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Oxon Hill, Maryland
  - Novo Nordisk Investigational Site, Flint, Michigan
  - Novo Nordisk Investigational Site, Billings, Montana
  - Novo Nordisk Investigational Site, Henderson, Nevada
  - Novo Nordisk Investigational Site, Albuquerque, New Mexico
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Whiteville, North Carolina
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Mentor, Ohio
  - Novo Nordisk Investigational Site, Wadsworth, Ohio
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Murrells Inlet, South Carolina
  - Novo Nordisk Investigational Site, Myrtle Beach, South Carolina
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Corpus Christi, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Chesapeake, Virginia
  - Novo Nordisk Investigational Site, Renton, Washington
- Argentina (3):
  - Novo Nordisk Investigational Site, CABA
  - Novo Nordisk Investigational Site, Corrientes
  - Novo Nordisk Investigational Site, Rosario
- Austria (3):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Saint Stefan
  - Novo Nordisk Investigational Site, Vienna
- Belgium (7):
  - Novo Nordisk Investigational Site, Bonheiden
  - Novo Nordisk Investigational Site, Boussu
  - Novo Nordisk Investigational Site, Brussels
  - Novo Nordisk Investigational Site, Edegem
  - Novo Nordisk Investigational Site, Ghent
  - Novo Nordisk Investigational Site, Leuven
  - Novo Nordisk Investigational Site, Liège
- Novo Nordisk Investigational Site, São Paulo, São Paulo, Brazil
- Egypt (2):
  - Novo Nordisk Investigational Site, Alexandria
  - Novo Nordisk Investigational Site, Cairo
- Norway (4):
  - Novo Nordisk Investigational Site, Hamar
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Stavanger
  - Novo Nordisk Investigational Site, Trondheim
- South Korea (5):
  - Novo Nordisk Investigational Site, Gangwon-do
  - Novo Nordisk Investigational Site, Gyeonggi-do
  - Novo Nordisk Investigational Site, Pusan
  - Novo Nordisk Investigational Site, Seoul
  - Novo Nordisk Investigational Site, Suwon
- Switzerland (7):
  - Novo Nordisk Investigational Site, Bern
  - Novo Nordisk Investigational Site, Einsiedeln
  - Novo Nordisk Investigational Site, Geneva
  - Novo Nordisk Investigational Site, Lucerne
  - Novo Nordisk Investigational Site, Olten
  - Novo Nordisk Investigational Site, Sankt Gallen
  - Novo Nordisk Investigational Site, Winterthur
- Turkey (Türkiye) (5):
  - Novo Nordisk Investigational Site, Adana
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Rize

IPD SHARING:
Plan to Share IPD: Yes
According to Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Result] Pieber TR, Bode B, Mertens A, Cho YM, Christiansen E, Hertz CL, Wallenstein SOR, Buse JB; PIONEER 7 investigators. Efficacy and safety of oral semaglutide with flexible dose adjustment versus sitagliptin in type 2 diabetes (PIONEER 7): a multicentre, open-label, randomised, phase 3a trial. Lancet Diabetes Endocrinol. 2019 Jul;7(7):528-539. doi: 10.1016/S2213-8587(19)30194-9. Epub 2019 Jun 9. PMID 31189520
- [Result] Buse JB, Bode BW, Mertens A, Cho YM, Christiansen E, Hertz CL, Nielsen MA, Pieber TR; PIONEER 7 investigators. Long-term efficacy and safety of oral semaglutide and the effect of switching from sitagliptin to oral semaglutide in patients with type 2 diabetes: a 52-week, randomized, open-label extension of the PIONEER 7 trial. BMJ Open Diabetes Res Care. 2020 Dec;8(2):e001649. doi: 10.1136/bmjdrc-2020-001649. PMID 33318068
- [Result] Aroda VR, Bauer R, Christiansen E, Haluzik M, Kallenbach K, Montanya E, Rosenstock J, Meier JJ. Efficacy and safety of oral semaglutide by subgroups of patient characteristics in the PIONEER phase 3 programme. Diabetes Obes Metab. 2022 Jul;24(7):1338-1350. doi: 10.1111/dom.14710. Epub 2022 May 9. PMID 35373893
- [Derived] Pratley RE, Crowley MJ, Gislum M, Hertz CL, Jensen TB, Khunti K, Mosenzon O, Buse JB. Oral Semaglutide Reduces HbA1c and Body Weight in Patients with Type 2 Diabetes Regardless of Background Glucose-Lowering Medication: PIONEER Subgroup Analyses. Diabetes Ther. 2021 Apr;12(4):1099-1116. doi: 10.1007/s13300-020-00994-9. Epub 2021 Mar 4. PMID 33660198
- [Derived] Husain M, Bain SC, Holst AG, Mark T, Rasmussen S, Lingvay I. Effects of semaglutide on risk of cardiovascular events across a continuum of cardiovascular risk: combined post hoc analysis of the SUSTAIN and PIONEER trials. Cardiovasc Diabetol. 2020 Sep 30;19(1):156. doi: 10.1186/s12933-020-01106-4. PMID 32998732
- [Derived] Thethi TK, Pratley R, Meier JJ. Efficacy, safety and cardiovascular outcomes of once-daily oral semaglutide in patients with type 2 diabetes: The PIONEER programme. Diabetes Obes Metab. 2020 Aug;22(8):1263-1277. doi: 10.1111/dom.14054. Epub 2020 May 13. PMID 32267058
- [Derived] Husain M, Bain SC, Jeppesen OK, Lingvay I, Sorrig R, Treppendahl MB, Vilsboll T. Semaglutide (SUSTAIN and PIONEER) reduces cardiovascular events in type 2 diabetes across varying cardiovascular risk. Diabetes Obes Metab. 2020 Mar;22(3):442-451. doi: 10.1111/dom.13955. Epub 2020 Feb 5. PMID 31903692
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The main phase of the trial was conducted at 77 sites in 10 countries, and the extension phase (Switch) at 71 sites in 9 countries, as follows (main phase/extension phase): Argentina (3/3), Austria (3/3), Belgium (7/7), Brazil (2/0), Egypt (4/4), Norway (4/4), South Korea (7/7), Switzerland (8/5), Turkey (8/8), and United States (31/30).
Pre-assignment Details: The trial consisted of two treatment periods: a 52-week main phase and a 52-week extension phase. In Switch, participants were allowed to re-randomise from sitagliptin to oral semaglutide. Sustainability included results for participants who received oral semaglutide during main + extension phase.
Groups:
- Oral Semaglutide Flex: Participants were to receive oral semaglutide tablets once daily from week 0 to week 52 (main phase): 3 milligrams (mg) for the first 8 weeks, 3 or 7 mg for next 8 weeks followed by 3, 7 or 14 mg for the remaining treatment period. Participants who were still on treatment at week 52 were allowed to continue on oral semaglutide in the extension phase (week 53 to week 104). Participants were to continue their anti-diabetic background medication (metformin, sulphonylurea, thiazolidinedione or sodium-glucose co-transporter 2 inhibitors) throughout the trial.
- Sitagliptin 100 mg- Main Phase: Participants were to receive 100 mg sitagliptin tablet once daily for 52 weeks (main phase). Participants were to continue their anti-diabetic background medication (metformin, sulphonylurea, thiazolidinedione or sodium-glucose co-transporter 2 inhibitors) throughout the trial (week 0 to week 52).
- Oral Semaglutide Flex- Switch: Participants who were still on sitagliptin 100 mg treatment at week 52 (end of main phase) were re-randomised to receive oral semaglutide tablets once daily from week 53 to week 104 (extension phase): 3 mg for the first 8 weeks, 3 or 7 mg for next 8 weeks followed by 3, 7 or 14 mg for the remaining treatment period. Participants were to continue their anti-diabetic background medication (metformin, sulphonylurea, thiazolidinedione or sodium-glucose co-transporter 2 inhibitors) throughout the trial (week 53 to week 104).
- Sitagliptin 100 mg- Switch: Participants who were still on sitagliptin 100 mg treatment at week 52 (end of main phase) were re-randomised to continue sitagliptin in the extension phase (week 53 to week 104). Participants were to continue their anti-diabetic background medication (metformin, sulphonylurea, thiazolidinedione or sodium-glucose co-transporter 2 inhibitors) throughout the trial (week 53 to week 104).
Period: Main Phase: 0 - 52 Weeks
Arm/Group | Oral Semaglutide Flex | Sitagliptin 100 mg- Main Phase | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Started | 253 | 251 | 0 | 0
Exposed | 253 | 250 | 0 | 0
Full Analysis Set (FAS) | 253 | 251 | 0 | 0
Safety Analysis Set (SAS) | 253 | 250 | 0 | 0
Completed | 241 | 244 | 0 | 0
Not Completed | 12 | 7 | 0 | 0
Not completed — Lost to Follow-up | 7 | 4 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 1 | 0 | 0
Not completed — Death | 0 | 2 | 0 | 0
Period: Extension Phase: 53 - 104 Weeks
Arm/Group | Oral Semaglutide Flex | Sitagliptin 100 mg- Main Phase | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Started | 185 (Participants who had provided consent to continue in the extension phase started in this period.) | 0 | 100 (Participants who had provided consent to continue in the extension phase started in this period.) | 98 (Participants who had provided consent to continue in the extension phase started in this period.)
Exposed | 184 | 0 | 100 | 97
Completed | 182 | 0 | 99 | 98
Not Completed | 3 | 0 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised participants. Baseline characteristics were presented for the participants who started in the Main phase of trial.
Groups:
- Sitagliptin 100 mg: Participants were to receive 100 mg sitagliptin tablet once daily for 52 weeks (main phase). Participants who were still on treatment at week 52 were re-randomised to continue sitagliptin in the extension phase (week 53 to week 104). Participants were to continue their anti-diabetic background medication (metformin, sulphonylurea, thiazolidinedione or sodium-glucose co-transporter 2 inhibitors) throughout the trial.
- Total: Total of all reporting groups
Arm/Group | Oral Semaglutide Flex | Sitagliptin 100 mg | Total
Number analyzed (Participants) | 253 | 251 | 504
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57 (10) | 58 (10) | 57 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 111 | 219
  Male | 145 | 140 | 285
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48 | 57 | 105
  Not Hispanic or Latino | 205 | 194 | 399
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 195 | 186 | 381
  Race: Black or African American | 22 | 25 | 47
  Race: Asian | 34 | 38 | 72
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  Race: Other | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Achieve HbA1c <7.0% (53 mmol/Mol) ADA Target (Yes/no)
Description: Participants who achieved HbA1c <7.0% (American Diabetes Association (ADA) target) (yes/no), was evaluated at week 52. The endpoint was evaluated based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product. The endpoint was also evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication and/or premature trial product discontinuation.
Time Frame: Week 52
Population: Overall number of participants analyzed = full analysis set (FAS) which comprised all randomised participants. Number Analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Groups:
- Oral Semaglutide Flex- Main Phase: Participants were to receive oral semaglutide tablets once daily from week 0 to week 52 (main phase): 3 milligrams (mg) for the first 8 weeks, 3 or 7 mg for next 8 weeks followed by 3, 7 or 14 mg for the remaining treatment period. Participants were to continue their anti-diabetic background medication (metformin, sulphonylurea, thiazolidinedione or sodium-glucose co-transporter 2 inhibitors) throughout the trial (week 0 to week 52).
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 253 | 251
Participants
  In-trial: number analyzed (Participants) | 230 | 238
  In-trial: Yes | 134 | 60
  In-trial: No | 96 | 178
  On-treatment without rescue medication: number analyzed (Participants) | 196 | 184
  On-treatment without rescue medication: Yes | 123 | 52
  On-treatment without rescue medication: No | 73 | 132
Statistical Analysis 1: Comparison: Oral Semaglutide Flex- Main Phase vs Sitagliptin 100 mg- Main Phase; The analysis was based on a pattern mixture model using multiple imputation to handle missing week 52 data, assuming that data were missing at random within the groups used for imputation. The imputed data sets were analysed using a logistic regression model with treatment, strata, and region as categorical fixed effects and baseline HbA1c value as covariate for each of the 1000 imputed complete datasets, and pooled by Rubin's rule to draw inference; Test type: Superiority — This hypothesis was controlled for multiplicity. Results are based on the data from the in-trial observation period. The estimated treatment effect includes the effect of any rescue medication and any effect after premature trial product discontinuation (treatment policy estimand); p < 0.0001, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from 1; Odds Ratio (OR) = 4.40, 95% CI 2-sided [2.89 to 6.70] — Oral Semaglutide flex / Sitagliptin 100 mg
Statistical Analysis 2: Comparison: Oral Semaglutide Flex- Main Phase vs Sitagliptin 100 mg- Main Phase; The analysis was based on multiple imputation, imputing sequentially using post-baseline measurements up to and including week 52. The imputed data sets were analysed using a logistic regression model with treatment, strata, and region as categorical fixed effects and baseline HbA1c value as covariate for each of the 1000 imputed complete datasets, and pooled by Rubin's rule to draw inference; Test type: Superiority — This hypothesis was not controlled for multiplicity. Results are based on the data from the on-treatment without rescue medication observation period. The estimated treatment effect excludes the effect of any rescue medication and any effect after premature trial product discontinuation (hypothetical estimand); p < 0.0001, Regression, Logistic — Unadjusted two-sided p-value for test of no difference from 1; Odds Ratio (OR) = 5.54, 95% CI 2-sided [3.54 to 8.68] — Oral Semaglutide flex / Sitagliptin 100 mg

2. Secondary Outcome: Change in Body Weight
Description: Change from baseline (week 0) in body weight was evaluated at week 52. The endpoint was evaluated based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product. The endpoint was also evaluated based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication and/or premature trial product discontinuation.
Time Frame: Week 0, week 52
Population: Overall number of participants analyzed = FAS which comprised all randomised participants. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Kilogram (Kg)
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 253 | 251
Kilogram (Kg)
  In-trial: number analyzed (Participants) | 233 | 239
  In-trial | -2.7 (3.9) | -0.7 (3.5)
  On-treatment without rescue medication: number analyzed (Participants) | 198 | 188
  On-treatment without rescue medication | -2.9 (4.0) | -0.9 (3.6)
Statistical Analysis 1: Comparison: Oral Semaglutide Flex- Main Phase vs Sitagliptin 100 mg- Main Phase; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Pattern mixture model — Unadjusted two-sided p-value for test of no difference from 0; Treatment difference = -1.9, 95% CI 2-sided [-2.6 to -1.2] — Oral semaglutide flex - Sitagliptin 100 mg
Statistical Analysis 2: Comparison: Oral Semaglutide Flex- Main Phase vs Sitagliptin 100 mg- Main Phase; The analysis was based on a Mixed model for repeated measurements (MMRM) that assumed data to be missing at random. As dependent variables, the MMRM model included all post-baseline values collected at scheduled visits up to and including week 52. The independent effects were treatment, strata and region as categorical fixed effects and the baseline HbA1c value as a covariate, all nested within visit, and an unstructured residual covariance matrix; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.0001, Mixed model for repeated measurements — Unadjusted two-sided p-value for test of no difference from 0; Treatment difference = -2.2, 95% CI 2-sided [-2.9 to -1.5] — Oral semaglutide flex - Sitagliptin 100 mg

3. Secondary Outcome: Change in HbA1c
Description: Change from baseline (week 0) in HbA1c was evaluated at week 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 230 | 238
Percentage of HbA1c | -1.3 (0.9) | -0.8 (1.0)

4. Secondary Outcome: Change in FPG
Description: Change from baseline (week 0) in fasting plasma glucose (FPG) was evaluated at week 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 229 | 232
Millimoles per liter (mmol/L) | -2.41 (2.35) | -1.39 (3.13)

5. Secondary Outcome: Change in Body Weight (%)
Description: Relative change from baseline (week 0) in body weight (kg) was evaluated at week 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 233 | 239
Percentage change | -2.99 (4.42) | -0.76 (3.91)

6. Secondary Outcome: Change in BMI
Description: Change from baseline (week 0) in body mass index (BMI) was evaluated at week 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, Week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Kilograms per square meter (kg/m^2)
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 233 | 239
Kilograms per square meter (kg/m^2) | -1.0 (1.5) | -0.3 (1.3)

7. Secondary Outcome: Change in Waist Circumference
Description: Change from baseline (week 0) in waist circumference was evaluated at week 52. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 231 | 237
Centimeters (cm) | -2.6 (5.3) | -0.7 (5.1)

8. Secondary Outcome: Change in Total Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in total cholesterol (mmol/L) at week 52 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, Week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 226 | 234
Ratio of total cholesterol | 0.96 (19.3) | 1.01 (16.2)

9. Secondary Outcome: Change in LDL Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in low-density lipoprotein (LDL) cholesterol (mmol/L) at week 52 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 226 | 233
Ratio of LDL cholesterol | 0.97 (31.8) | 1.03 (27.2)

10. Secondary Outcome: Change in HDL Cholesterol (Ratio to Baseline)
Description: Change from baseline (week 0) in high-density lipoprotein (HDL) cholesterol (mmol/L) at weeks 26, 52 and 78 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 226 | 233
Ratio of HDL cholesterol | 1.00 (14.0) | 1.02 (16.5)

11. Secondary Outcome: Change in Triglycerides (Ratio to Baseline)
Description: Change from baseline (week 0) in triglycerides (mmol/L) at week 52 is presented as ratio to baseline. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 226 | 233
Ratio of triglycerides | 0.89 (38.2) | 0.91 (43.1)

12. Secondary Outcome: Change in SF-36v2 (Acute Version) Health Survey: Scores From the 8 Domains, the Physical Component Summary (PCS) and the Mental Component Summary (MCS)
Description: SF-36 is a 36-item patient-reported survey of patient health that measures the participant's overall health-related quality of life (HRQoL). SF-36v2™ (acute version) questionnaire measured eight domains of functional health and well-being as well as two component summary scores (physical component summary (PCS) and mental component summary (MCS)). The 0-100 scale scores (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. In the metric of norm-based scores, 50 and 10 corresponds to the mean and standard deviation respectively of the 2009 U.S. general population. Change from baseline (week 0) in the domain scores and component summary (PCS and MCS) scores were evaluated at week 52. A positive change score indicates an improvement since baseline. Results are based on the data from the in-trial observation period.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 253 | 251
Score on a scale
  Physical functioning: number analyzed (Participants) | 230 | 239
  Physical functioning | 1.54 (7.92) | -0.03 (7.16)
  Role physical: number analyzed (Participants) | 231 | 239
  Role physical | 0.40 (7.82) | 0.13 (8.38)
  Bodily pain: number analyzed (Participants) | 231 | 239
  Bodily pain | 1.09 (9.01) | 1.20 (8.72)
  General health: number analyzed (Participants) | 231 | 239
  General health | 1.83 (7.65) | 1.62 (6.71)
  Vitality: number analyzed (Participants) | 229 | 239
  Vitality | 1.07 (8.16) | 0.51 (7.28)
  Social functioning: number analyzed (Participants) | 231 | 239
  Social functioning | 0.38 (9.00) | 0.41 (7.86)
  Role emotional: number analyzed (Participants) | 231 | 239
  Role emotional | -0.91 (11.71) | -0.54 (10.58)
  Mental health: number analyzed (Participants) | 229 | 239
  Mental health | 1.21 (8.54) | 0.86 (7.97)
  PCS: number analyzed (Participants) | 229 | 239
  PCS | 1.51 (6.39) | 0.74 (5.81)
  MCS: number analyzed (Participants) | 229 | 239
  MCS | 0.01 (8.75) | 0.26 (7.67)

13. Secondary Outcome: Change in DTSQ
Description: Change from baseline (week 0) in diabetes treatment satisfaction questionnaire - status (DTSQs) was evaluated at week 52. The DTSQs items are scored on a 7-point graded response scale ranging from 6 to 0. Higher scores indicate higher levels of treatment satisfaction for DTSQs items 1, 4 -8. For items 2 and 3 a higher score indicates a higher patient perceived experience of high blood sugars and low blood sugars, respectively. Thus, lower scores indicate a perception of blood glucose levels being "none of the time" unacceptably high (item 2) or low (item 3). The domain score of total treatment satisfaction (total treatment satisfaction score) was computed by adding the six items scores 1, 4-8. The score ranges 0-36. A higher treatment satisfaction score indicates a higher level of treatment satisfaction. Results are based on the data from the in-trial observation period.
Time Frame: Week 0, Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 253 | 251
Score on a scale
  1) Satisfaction with treatment: number analyzed (Participants) | 230 | 239
  1) Satisfaction with treatment | 1.09 (1.61) | 0.92 (1.65)
  2) Feeling of unacceptably high blood sugars: number analyzed (Participants) | 231 | 239
  2) Feeling of unacceptably high blood sugars | -1.58 (2.13) | -1.14 (2.13)
  3) Feeling of unacceptably low blood sugars: number analyzed (Participants) | 228 | 238
  3) Feeling of unacceptably low blood sugars | -0.15 (1.70) | -0.24 (1.99)
  4) Convenience of treatment: number analyzed (Participants) | 229 | 234
  4) Convenience of treatment | 0.82 (1.54) | 0.59 (1.48)
  5) Flexibility of current treatment: number analyzed (Participants) | 231 | 239
  5) Flexibility of current treatment | 0.80 (1.58) | 0.68 (1.51)
  6) Satisfaction with understanding of diabetes: number analyzed (Participants) | 231 | 239
  6) Satisfaction with understanding of diabetes | 0.77 (1.51) | 0.77 (1.71)
  7) Recommending treatment to others: number analyzed (Participants) | 231 | 237
  7) Recommending treatment to others | 0.88 (1.54) | 0.79 (1.46)
  8) Satisfaction to continue with present treatment: number analyzed (Participants) | 229 | 238
  8) Satisfaction to continue with present treatment | 1.03 (1.66) | 0.95 (1.88)
  Total treatment satisfaction score: number analyzed (Participants) | 231 | 239
  Total treatment satisfaction score | 5.39 (6.84) | 4.70 (7.23)

14. Secondary Outcome: Participants Who Achieve HbA1c ≤6.5% (48 mmol/Mol) AACE Target (Yes/no)
Description: Participants who achieved HbA1c less than or equal to 6.5% (American Association of Clinical Endocrinologists (AACE) target) (yes/no) at week 52 is presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 230 | 238
Participants
  Yes | 76 | 29
  No | 154 | 209

15. Secondary Outcome: Participants Who Achieve Weight Loss ≥5% (Yes/no)
Description: Participants who achieved weight loss more than or equal to 5% of their baseline body weight (yes/no) at weeks 52 is presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 233 | 239
Participants
  Yes | 63 | 29
  No | 170 | 210

16. Secondary Outcome: Participants Who Achieve Weight Loss ≥10% (Yes/no)
Description: Participants who achieved weight loss more than or equal to 10% of their baseline body weight (yes/no) at week 52 is presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 233 | 239
Participants
  Yes | 15 | 5
  No | 218 | 234

17. Secondary Outcome: Participants Who Achieve HbA1c <7.0 % (53 mmol/Mol) Without Hypoglycaemia (Severe or BG Confirmed Symptomatic Hypoglycaemia) and no Weight Gain (Yes/no)
Description: Participants who achieved HbA1c less than 7.0 % without severe or blood glucose (BG) confirmed symptomatic hypoglycaemia and without weight gain (yes/no) at week 52 is presented. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia was defined as an episode with plasma glucose value <3.1 mmol/L with symptoms consistent with hypoglycaemia. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 230 | 238
Participants
  Yes | 104 | 35
  No | 126 | 203

18. Secondary Outcome: Participants Who Achieve HbA1c Reduction ≥1% (10.9 mmol/Mol) and Weight Loss ≥3% (Yes/no)
Description: Participants who achieved HbA1c reduction more than or equal to 1% of their baseline HbA1c and weight loss of more than or equal to 3% of their baseline body weight (yes/no) at week 52 is presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 230 | 238
Participants
  Yes | 80 | 25
  No | 150 | 213

19. Secondary Outcome: Time to Rescue Medication
Description: Presented results are the number of participants who had taken rescue medication anytime during the periods, from week 0 to week 52. Rescue medication was defined as any new anti-diabetic medication used as add-on to trial product and used for more than 21 days with the initiation at or after randomisation (week 0) and before last day on trial product, and/or intensification of anti-diabetic medication (a more than 20% increase in dose relative to baseline) for more than 21 days with the intensification at or after randomisation and before last day on trial product. Results are based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication and/or premature trial product discontinuation.
Time Frame: Weeks 0-52
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 253 | 251
Participants | 8 | 40
Statistical Analysis 1: Comparison: Oral Semaglutide Flex- Main Phase vs Sitagliptin 100 mg- Main Phase; Time to initiation of rescue medication was analysed using a Cox proportional hazards model with treatment, strata, and region as categorical fixed effects and baseline HbA1c as covariate. Censoring time was one day before last day on trial product; Test type: Superiority — This hypothesis was not controlled for multiplicity; p < 0.0001, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.18, 95% CI 2-sided [0.09 to 0.39] — Oral semaglutide flex / Sitagliptin 100 mg

20. Secondary Outcome: Time to Additional Anti-diabetic Medication
Description: Presented results are the number of participants who had taken additional anti-diabetic medication anytime during the period from week 0 to week 52. Additional anti-diabetic medication was defined as any new anti-diabetic medication used for more than 21 days with the initiation at or after randomisation (week 0) and before (planned) end-of-treatment (week 52), and/or intensification of anti-diabetic medication (a more than 20% increase in dose relative to baseline) for more than 21 days with the intensification at or after randomisation and before (planned) end-of-treatment. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Weeks 0-52
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 253 | 251
Participants | 22 | 47
Statistical Analysis 1: Comparison: Oral Semaglutide Flex- Main Phase vs Sitagliptin 100 mg- Main Phase; Time to initiation of additional anti-diabetic medication was analysed using a Cox proportional hazards model with treatment, strata, and region as categorical fixed effects and baseline HbA1c as covariate. Censoring time was one day before planned end of treatment; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0175, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.37 to 0.91] — Oral Semaglutide flex / Sitagliptin 100 mg

21. Secondary Outcome: Number of TEAEs During Exposure to Trial Product
Description: Treatment emergent adverse events (TEAEs) were recorded from week 0 to week 57 (52-week treatment period for participants who continued in the extension phase; 52-week treatment period plus the 5-week follow-up period for participants who did not continue in the extension phase). Adverse events (AEs) with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period: Time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0-57
Population: Overall number of participants analyzed = safety analysis set (SAS) which comprised all randomised participants who received at least one dose of trial product.
Measure: Number; unit: Events
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 253 | 250
Events | 768 | 519

22. Secondary Outcome: Number of Treatment-emergent Severe or BG-confirmed Symptomatic Hypoglycaemic Episodes
Description: Treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes were recorded during weeks 0-57 (52-week treatment period for participants who continued in the extension phase; 52-week treatment period plus the 5-week follow-up period for participants who did not continue in the extension phase). Hypoglycaemic episodes with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period was defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia: Confirmed by a glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: Week 0-57
Population: Overall number of participants analyzed = SAS which comprised all randomised participants who received at least one dose of trial product.
Measure: Number; unit: Episodes
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 253 | 250
Episodes | 34 | 22

23. Secondary Outcome: Paticipants With Treatment-emergent Severe or BG-confirmed Symptomatic Hypoglycaemic Episodes (Yes/no)
Description: as for outcome 22
Time Frame: Week 0-57
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 253 | 250
Participants | 14 | 14

24. Secondary Outcome: Change in Amylase (Ratio to Baseline)
Description: Change from baseline (week 0) in biochemical parameter- amylase (units per liter [U/L]) to week 52 is presented as ratio to baseline. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, Week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of amylase
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 201 | 225
Ratio of amylase | 1.14 (25.5) | 1.08 (26.3)

25. Secondary Outcome: Change in Lipase (Ratio to Baseline)
Description: Change from baseline (week 0) in lipase (U/L) to week 52 is presented as ratio to baseline. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, Week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of lipase
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 201 | 225
Ratio of lipase | 1.24 (55.2) | 1.13 (55.3)

26. Secondary Outcome: Change in Pulse Rate
Description: Change from baseline (week 0) in pulse rate was evaluated at week 52. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 206 | 225
Beats per minute | 3 (9) | 0 (10)

27. Secondary Outcome: Change in Blood Pressure (Systolic and Diastolic Blood Pressure)
Description: Change from baseline (week 0) in systolic blood pressure (SBP) and diastolic blood pressure (DBP) was evaluated at week 52. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 52
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase
Number analyzed (Participants) | 206 | 225
Millimeters of mercury (mmHg)
  Systolic blood pressure | -3 (14) | -2 (15)
  Diastolic blood pressure | -0 (9) | -1 (10)

28. Secondary Outcome: Change in HbA1c- Switch
Description: Change from week 52 in HbA1c was evaluated at week 104. Results are based on the data from the in-trial observation period, which was the time period from when a participant was re-randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 52, week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Number analyzed (Participants) | 92 | 96
Percentage of HbA1c | -0.2 (1.2) | 0.0 (1.0)

29. Secondary Outcome: Change in Body Weight- Switch
Description: Change from week 52 in body weight was evaluated at week 104. Results are based on the data from the in-trial observation period, which was the time period from when a participant was re-randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 52, week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Number analyzed (Participants) | 93 | 97
Kg | -2.6 (3.8) | -0.9 (5.4)

30. Secondary Outcome: Change in Body Weight (%)- Switch
Description: Relative change from week 52 in body weight (kg) was evaluated at week 104. Results are based on the data from the in-trial observation period, which was the time period from when a participant was re-randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 52, week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Number analyzed (Participants) | 93 | 97
Percentage change | -3.12 (4.50) | -0.70 (5.27)

31. Secondary Outcome: Change in FPG- Switch
Description: Change from week 52 in fasting plasma glucose (FPG) was evaluated at week 104. Results are based on the data from the in-trial observation period, which was the time period from when a participant was re-randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 52, week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Number analyzed (Participants) | 92 | 94
Millimoles per liter (mmol/L) | -0.35 (1.95) | 0.02 (2.31)

32. Secondary Outcome: Change in BMI- Switch
Description: Change from week 52 in body mass index (BMI) was evaluated at week 104. Results are based on the data from the in-trial observation period, which was the time period from when a participant was re-randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 52, Week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Number analyzed (Participants) | 93 | 97
kg/m^2 | -0.9 (1.4) | -0.3 (2.2)

33. Secondary Outcome: Change in Waist Circumference- Switch
Description: Change from week 52 in waist circumference was evaluated at week 104. Results are based on the data from the in-trial observation period, which was the time period from when a participant was re-randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 52, week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Number analyzed (Participants) | 93 | 97
Centimeters (cm) | -1.8 (4.3) | -0.9 (5.8)

34. Secondary Outcome: Participants Who Achieve HbA1c <7.0% (53 mmol/Mol) ADA Target (Yes/no)- Switch
Description: Participants who achieved HbA1c <7.0% (American Diabetes Association (ADA) target) (yes/no), was evaluated at week 104. The endpoint was evaluated based on the data from the in-trial observation period, which was the time period from when a participant was re-randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 104 (i.e., after 52 weeks of treatment in the extension phase)
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Number analyzed (Participants) | 92 | 96
Participants
  Yes | 44 | 26
  No | 48 | 70

35. Secondary Outcome: Participants Who Achieve HbA1c ≤6.5% (48 mmol/Mol) AACE Target (Yes/no)- Switch
Description: Participants who achieved HbA1c less than or equal to 6.5% (American Association of Clinical Endocrinologists (AACE) target) (yes/no) at week 104 is presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was re-randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 104 (i.e., after 52 weeks of treatment in the extension phase)
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Number analyzed (Participants) | 92 | 96
Participants
  Yes | 28 | 11
  No | 64 | 85

36. Secondary Outcome: Participants Who Achieve Weight Loss ≥5% (Yes/no)- Switch
Description: Participants who achieved weight loss more than or equal to 5% of their baseline body weight (yes/no) at weeks 104 is presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was re-randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 104 (i.e., after 52 weeks of treatment in the extension phase)
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Number analyzed (Participants) | 93 | 97
Participants
  Yes | 31 | 12
  No | 62 | 85

37. Secondary Outcome: Participants Who Achieve HbA1c <7.0% (53 mmol/Mol) Without Hypoglycaemia (Severe or BG Confirmed Symptomatic Hypoglycaemia) and no Weight Gain (Yes/no)- Switch
Description: Participants who achieved HbA1c less than 7.0% without severe or blood glucose (BG) confirmed symptomatic hypoglycaemia and without weight gain (yes/no) at week 104 is presented. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia was defined as an episode with plasma glucose value <3.1 mmol/L with symptoms consistent with hypoglycaemia. Results are based on the data from the in-trial observation period, which was the time period from when a participant was re-randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 104 (i.e., after 52 weeks of treatment in the extension phase)
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Number analyzed (Participants) | 92 | 96
Participants
  Yes | 36 | 18
  No | 56 | 78

38. Secondary Outcome: Participants Who Achieve HbA1c <7.0% (53 mmol/Mol) ADA Target and no Need for Rescue Medication (Yes/no)- Switch
Description: Participants who achieved HbA1c <7.0% (American Diabetes Association (ADA) target) and no need for rescue medication (yes/no), was evaluated at week 104. Results are based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication and/or premature trial product discontinuation.
Time Frame: Week 104 (i.e., after 52 weeks of treatment in the extension phase)
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Number analyzed (Participants) | 92 | 96
Participants | 41 | 23

39. Secondary Outcome: Time to Additional Anti-diabetic Medication- Switch
Description: Presented results are the number of participants who had taken additional anti-diabetic medication anytime during the period from week 53 to week 104. Additional anti-diabetic medication was defined as any new anti-diabetic medication used for more than 21 days with the initiation at or after re-randomisation (week 52) and before (planned) end-of-treatment (week 104), and/or intensification of anti-diabetic medication (a more than 20% increase in dose relative to baseline) for more than 21 days with the intensification at or after randomisation and before (planned) end-of-treatment. Results are based on the data from the in-trial observation period, which was the time period from when a participant was re-randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Weeks 53-104
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Number analyzed (Participants) | 100 | 98
Participants | 15 | 26
Statistical Analysis 1: Comparison: Oral Semaglutide Flex- Switch vs Sitagliptin 100 mg- Switch; [analysis description as in outcome 20, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.4381, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.39 to 1.50] — Oral Semaglutide flex- Switch / Sitagliptin 100 mg- Switch

40. Secondary Outcome: Time to Rescue Medication- Switch
Description: Presented results are the number of participants who had taken rescue medication anytime during the periods, from week 53 to week 104. Rescue medication was defined as any new anti-diabetic medication used as add-on to trial product and used for more than 21 days with the initiation at or after re-randomisation (week 52) and before last day on trial product, and/or intensification of anti-diabetic medication (a more than 20% increase in dose relative to baseline) for more than 21 days with the intensification at or after randomisation and before last day on trial product. Results are based on the data from the on-treatment without rescue medication observation period, which was the time period when a participant was on treatment with trial product, excluding any period after initiation of rescue medication and/or premature trial product discontinuation.
Time Frame: Weeks 53-104
Population: Overall number of participants analyzed = FAS which comprised all randomised participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Number analyzed (Participants) | 100 | 98
Participants | 9 | 23
Statistical Analysis 1: Comparison: Oral Semaglutide Flex- Switch vs Sitagliptin 100 mg- Switch; [analysis description as in outcome 19, analysis 1]; Test type: Superiority — This hypothesis was not controlled for multiplicity; p = 0.0790, Regression, Cox — Unadjusted two-sided p-value for test of no difference from 1; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.20 to 1.09] — Oral semaglutide flex- Switch / Sitagliptin 100 mg- Switch

41. Secondary Outcome: Number of TEAEs During Exposure to Trial Product- Switch
Description: Treatment emergent adverse events (TEAEs) were recorded from week 53 to week 109. Adverse events (AEs) with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period: Time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 53-109
Population: as for outcome 21
Measure: Number; unit: Events
Arm/Group | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Number analyzed (Participants) | 100 | 97
Events | 267 | 225

42. Secondary Outcome: Change in Amylase (Ratio to Baseline)- Switch
Description: Change from week 52 in biochemical parameter- amylase (U/L) to week 104 is presented as ratio to baseline. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 52, Week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of amylase
Arm/Group | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Number analyzed (Participants) | 84 | 92
Ratio of amylase | 1.09 (22.9) | 1.00 (26.6)

43. Secondary Outcome: Change in Lipase (Ratio to Baseline)- Switch
Description: Change from week 52 in lipase (U/L) to week 104 is presented as ratio to baseline. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 52, Week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of lipase
Arm/Group | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Number analyzed (Participants) | 84 | 92
Ratio of lipase | 1.13 (46.7) | 0.92 (54.9)

44. Secondary Outcome: Change in Pulse Rate- Switch
Description: Change from week 52 in pulse rate was evaluated at week 104. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 52, week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Number analyzed (Participants) | 87 | 93
Beats per minute | 1 (9) | -0 (10)

45. Secondary Outcome: Change in Blood Pressure (Systolic and Diastolic Blood Pressure)- Switch
Description: Change from week 52 in systolic blood pressure (SBP) and diastolic blood pressure (DBP) was evaluated at week 104. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 52, week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Number analyzed (Participants) | 87 | 93
Millimeters of mercury (mmHg)
  Systolic blood pressure | -3 (15) | 2 (15)
  Diastolic blood pressure | -1 (10) | -0 (10)

46. Secondary Outcome: Number of Treatment-emergent Severe or BG-confirmed Symptomatic Hypoglycaemic Episodes- Switch
Description: Treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes were recorded during weeks 53 to 109. Hypoglycaemic episodes with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period was defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia: Confirmed by a glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: Week 53-109
Population: as for outcome 22
Measure: Number; unit: Episodes
Arm/Group | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Number analyzed (Participants) | 100 | 97
Episodes | 2 | 12

47. Secondary Outcome: Paticipants With Treatment-emergent Severe or BG-confirmed Symptomatic Hypoglycaemic Episodes (Yes/no)- Switch
Description: Number of participants with treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes were recorded during weeks 53 to 109. Hypoglycaemic episodes with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period was defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia: Confirmed by a glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: Week 53-109
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Number analyzed (Participants) | 100 | 97
Participants | 2 | 4

48. Secondary Outcome: Change in SF-36v2 (Acute Version) Health Survey: Scores From the 8 Domains, the Physical Component Summary (PCS) and the Mental Component Summary (MCS)- Switch
Description: SF-36 is a 36-item patient-reported survey of patient health that measures the participant's overall health-related quality of life (HRQoL). SF-36v2™ (acute version) questionnaire measured eight domains of functional health and well-being as well as two component summary scores (physical component summary (PCS) and mental component summary (MCS)). The 0-100 scale scores (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. In the metric of norm-based scores, 50 and 10 corresponds to the mean and standard deviation respectively of the 2009 U.S. general population. Change from week 52 in the domain scores and component summary (PCS and MCS) scores were evaluated at week 104. A positive change score indicates an improvement since week 52. Results are based on the data from the in-trial observation period.
Time Frame: Week 52, week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Number analyzed (Participants) | 93 | 97
Score on a scale
  Physical functioning | 1.14 (8.55) | -0.97 (6.71)
  Role physical | 1.37 (7.68) | -0.22 (7.61)
  Bodily pain | -0.18 (7.22) | -0.30 (7.06)
  General health | 0.69 (6.74) | 0.53 (6.59)
  Vitality | -0.18 (6.91) | -0.15 (7.32)
  Social functioning | 0.21 (7.36) | 0.10 (6.54)
  Role emotional | 1.72 (9.61) | -0.39 (8.79)
  Mental health | 0.37 (6.68) | 0.20 (6.46)
  PCS | 0.66 (6.06) | -0.43 (5.36)
  MCS | 0.52 (7.21) | 0.19 (6.46)

49. Secondary Outcome: Change in DTSQ- Switch
Description: Change from week 52 in diabetes treatment satisfaction questionnaire - status (DTSQs) was evaluated at week 104. The DTSQs items are scored on a 7-point graded response scale ranging from 6 to 0. Higher scores indicate higher levels of treatment satisfaction for DTSQs items 1, 4 -8. For items 2 and 3 a higher score indicates a higher patient perceived experience of high blood sugars and low blood sugars, respectively. Thus, lower scores indicate a perception of blood glucose levels being "none of the time" unacceptably high (item 2) or low (item 3). The domain score of total treatment satisfaction (total treatment satisfaction score) was computed by adding the six items scores 1, 4-8. The score ranges 0-36. A higher treatment satisfaction score indicates a higher level of treatment satisfaction. Results are based on the data from the in-trial observation period.
Time Frame: Week 52, week 104
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
Number analyzed (Participants) | 100 | 98
Score on a scale
  1) Satisfaction with treatment: number analyzed (Participants) | 93 | 97
  1) Satisfaction with treatment | 0.06 (1.06) | -0.24 (1.43)
  2) Feeling of unacceptably high blood sugars: number analyzed (Participants) | 93 | 97
  2) Feeling of unacceptably high blood sugars | -0.32 (1.95) | 0.09 (2.04)
  3) Feeling of unacceptably low blood sugars: number analyzed (Participants) | 93 | 97
  3) Feeling of unacceptably low blood sugars | 0.02 (1.63) | 0.23 (1.94)
  4) Convenience of treatment: number analyzed (Participants) | 92 | 94
  4) Convenience of treatment | 0.13 (1.18) | 0.13 (1.16)
  5) Flexibility of current treatment: number analyzed (Participants) | 93 | 97
  5) Flexibility of current treatment | 0.01 (1.19) | 0.06 (1.22)
  6) Satisfaction with understanding of diabetes: number analyzed (Participants) | 93 | 97
  6) Satisfaction with understanding of diabetes | 0.02 (1.38) | 0.04 (1.16)
  7) Recommending treatment to others: number analyzed (Participants) | 92 | 96
  7) Recommending treatment to others | 0.04 (1.04) | -0.05 (1.20)
  8) Satisfaction to continue with present treatment: number analyzed (Participants) | 92 | 97
  8) Satisfaction to continue with present treatment | -0.05 (1.07) | 0.00 (1.48)
  Total treatment satisfaction score: number analyzed (Participants) | 93 | 97
  Total treatment satisfaction score | 0.20 (5.14) | -0.06 (5.62)

50. Secondary Outcome: Change in HbA1c- Sustainability
Description: Change from baseline (week 0) in HbA1c was evaluated at week 104. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Groups:
- Oral Semaglutide Flex- Sustainability: Participants were to receive oral semaglutide tablets once daily for 104 weeks (week 0-52 in the main phase and week 53-104 in the extension phase): 3 mg for the first 8 weeks, 3 or 7 mg for next 8 weeks followed by 3, 7 or 14 mg for the remaining treatment period. Participants were to continue their anti-diabetic background medication (metformin, sulphonylurea, thiazolidinedione or sodium-glucose co-transporter 2 inhibitors) throughout the trial (week 0 to week 104).
Arm/Group | Oral Semaglutide Flex- Sustainability
Number analyzed (Participants) | 180
Percentage of HbA1c | -1.3 (1.0)

51. Secondary Outcome: Change in Body Weight (kg)- Sustainability
Description: Change from baseline (week 0) in body weight was evaluated at week 104. The endpoint was evaluated based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Oral Semaglutide Flex- Sustainability
Number analyzed (Participants) | 180
Kg | -3.7 (5.2)

52. Secondary Outcome: Change in Body Weight (%)- Sustainability
Description: Relative change from baseline (week 0) in body weight (kg) was evaluated at week 104. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Oral Semaglutide Flex- Sustainability
Number analyzed (Participants) | 180
Percentage change | -4.03 (5.75)

53. Secondary Outcome: Change in FPG- Sustainability
Description: Change from baseline (week 0) in fasting plasma glucose (FPG) was evaluated at week 104. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Oral Semaglutide Flex- Sustainability
Number analyzed (Participants) | 178
Millimoles per liter (mmol/L) | -39.4 (51.2)

54. Secondary Outcome: Change in BMI- Sustainability
Description: Change from baseline (week 0) in body mass index (BMI) was evaluated at week 104. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, Week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Oral Semaglutide Flex- Sustainability
Number analyzed (Participants) | 180
kg/m^2 | -1.3 (1.9)

55. Secondary Outcome: Change in Waist Circumference- Sustainability
Description: Change from baseline (week 0) in waist circumference was evaluated at week 104. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 0, week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Oral Semaglutide Flex- Sustainability
Number analyzed (Participants) | 178
cm | -2.5 (6.3)

56. Secondary Outcome: Participants Who Achieve HbA1c <7.0% (53 mmol/Mol) ADA Target (Yes/no)- Sustainability
Description: Participants who achieved HbA1c <7.0% (American Diabetes Association (ADA) target) (yes/no), was evaluated at week 104. The endpoint was evaluated based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide Flex- Sustainability
Number analyzed (Participants) | 180
Participants
  Yes | 101
  No | 79

57. Secondary Outcome: Participants Who Achieve HbA1c ≤6.5% (48 mmol/Mol) AACE Target (Yes/no)- Sustainability
Description: Participants who achieved HbA1c less than or equal to 6.5% (American Association of Clinical Endocrinologists (AACE) target) (yes/no) at week 104 is presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide Flex- Sustainability
Number analyzed (Participants) | 180
Participants
  Yes | 63
  No | 117

58. Secondary Outcome: Participants Who Achieve Weight Loss ≥5% (Yes/no)- Sustainability
Description: Participants who achieved weight loss more than or equal to 5% of their baseline body weight (yes/no) at weeks 104 is presented. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide Flex- Sustainability
Number analyzed (Participants) | 180
Participants
  Yes | 61
  No | 119

59. Secondary Outcome: Participants Who Achieve HbA1c <7.0 % (53 mmol/Mol) Without Hypoglycaemia (Severe or BG Confirmed Symptomatic Hypoglycaemia) and no Weight Gain (Yes/no)- Sustainability
Description: Participants who achieved HbA1c less than 7.0 % without severe or blood glucose (BG) confirmed symptomatic hypoglycaemia and without weight gain (yes/no) at week 104 is presented. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia was defined as an episode with plasma glucose value <3.1 mmol/L with symptoms consistent with hypoglycaemia. Results are based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide Flex- Sustainability
Number analyzed (Participants) | 180
Participants
  Yes | 73
  No | 107

60. Secondary Outcome: Participants Who Achieve HbA1c <7.0% (53 mmol/Mol) ADA Target or HbA1c Reduction ≥ 1%-Point (10.9 mmol/Mol) (Yes/no)- Sustainability
Description: Participants who achieved HbA1c <7.0% ADA target or HbA1c reduction ≥ 1%-point (10.9 mmol/mol) (yes/no), was evaluated at week 104. The endpoint was evaluated based on the data from the in-trial observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Time Frame: Week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide Flex- Sustainability
Number analyzed (Participants) | 180
Participants
  Yes | 126
  No | 54

61. Secondary Outcome: Number of TEAEs During Exposure to Trial Product- Sustainability
Description: Treatment emergent adverse events (TEAEs) were recorded from week 0 to week 109 ((104-week treatment period for participants who continued in the extension phase or 52-week treatment period for participants who did not continue in the extension phase) plus the 5-week follow-up period). Adverse events (AEs) with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period: Time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0-109
Population: as for outcome 22
Measure: Number; unit: Events
Arm/Group | Oral Semaglutide Flex- Sustainability
Number analyzed (Participants) | 253
Events | 1157

62. Secondary Outcome: Change in Amylase (Ratio to Baseline)- Sustainability
Description: Change from baseline (week 0) in biochemical parameter- amylase (units per liter [U/L]) to week 104 is presented as ratio to baseline. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of amylase
Arm/Group | Oral Semaglutide Flex- Sustainability
Number analyzed (Participants) | 167
Ratio of amylase | 1.13 (25.1)

63. Secondary Outcome: Change in Lipase (Ratio to Baseline)- Sustainability
Description: Change from baseline (week 0) in lipase (U/L) to week 104 is presented as ratio to baseline. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, Week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of lipase
Arm/Group | Oral Semaglutide Flex- Sustainability
Number analyzed (Participants) | 167
Ratio of lipase | 1.18 (58.0)

64. Secondary Outcome: Change in Pulse Rate- Sustainability
Description: Change from baseline (week 0) in pulse rate was evaluated at week 104. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Oral Semaglutide Flex- Sustainability
Number analyzed (Participants) | 176
Beats per minute | 2 (9)

65. Secondary Outcome: Change in Blood Pressure (Systolic and Diastolic Blood Pressure)- Sustainability
Description: Change from baseline (week 0) in systolic blood pressure (SBP) and diastolic blood pressure (DBP) was evaluated at week 104. Results are based on the data from the on-treatment observation period which was the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication.
Time Frame: Week 0, week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Oral Semaglutide Flex- Sustainability
Number analyzed (Participants) | 176
Millimeters of mercury (mmHg)
  Systolic blood pressure | -3 (14)
  Diastolic blood pressure | -1 (9)

66. Secondary Outcome: Number of Treatment-emergent Severe or BG-confirmed Symptomatic Hypoglycaemic Episodes)- Sustainability
Description: Treatment emergent severe or BG confirmed symptomatic hypoglycaemic episodes were recorded during weeks 0-109 ((104-week treatment period for participants who continued in the extension phase or 52-week treatment period for participants who did not continue in the extension phase) plus the 5-week follow-up period). Hypoglycaemic episodes with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period was defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia: Confirmed by a glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: Week 0-109
Population: as for outcome 22
Measure: Number; unit: Episodes
Arm/Group | Oral Semaglutide Flex- Sustainability
Number analyzed (Participants) | 253
Episodes | 45

67. Secondary Outcome: Paticipants With Treatment-emergent Severe or BG-confirmed Symptomatic Hypoglycaemic Episodes (Yes/no)- Sustainability
Description: Number of participants with treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes were recorded during weeks 0-109 ((104-week treatment period for participants who continued in the extension phase or 52-week treatment period for participants who did not continue in the extension phase) plus the 5-week follow-up period). Hypoglycaemic episodes with onset during the on-treatment observation period were considered treatment-emergent. On-treatment observation period was defined as the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication. Severe hypoglycaemia was defined as an episode requiring assistance of another person to actively administer carbohydrate or glucagon, or take other corrective actions. BG-confirmed symptomatic hypoglycaemia: Confirmed by a glucose value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: Week 0-109
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Semaglutide Flex- Sustainability
Number analyzed (Participants) | 253
Participants | 18

68. Secondary Outcome: Change in SF-36v2 (Acute Version) Health Survey: Scores From the 8 Domains, the Physical Component Summary (PCS) and the Mental Component Summary (MCS)- Sustainability
Description: Short form (SF)-36 is a 36-item patient-reported survey of patient health that measures the participant's overall health-related quality of life (HRQoL). SF-36v2™ (acute version) questionnaire measured eight domains of functional health and well-being as well as two component summary scores (physical component summary (PCS) and mental component summary (MCS)). The 0-100 scale scores (where higher scores indicated a better HRQoL) from the SF-36 were converted to norm-based scores to enable a direct interpretation in relation to the distribution of the scores in the 2009 U.S. general population. In the metric of norm-based scores, 50 and 10 corresponds to the mean and standard deviation respectively of the 2009 U.S. general population. Change from baseline (week 0) in the domain scores and component summary (PCS and MCS) scores were evaluated at week 104. A positive change score indicates an improvement since baseline. Results are based on the data from the in-trial observation period.
Time Frame: Week 0, week 104
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide Flex- Sustainability
Number analyzed (Participants) | 180
Score on a scale
  Physical functioning | 1.44 (8.48)
  Role physical | 0.22 (8.31)
  Bodily pain | 1.07 (9.72)
  General health | 1.98 (8.01)
  Vitality | 0.97 (8.49)
  Social functioning | -0.11 (8.14)
  Role emotional | -0.04 (10.49)
  Mental health | 1.05 (8.25)
  PCS | 1.33 (6.96)
  MCS | 0.20 (8.34)

69. Secondary Outcome: Change in DTSQ- Sustainability
Description: Change from week 0 in diabetes treatment satisfaction questionnaire - status (DTSQs) was evaluated at week 104. The DTSQs items are scored on a 7-point graded response scale ranging from 6 to 0. Higher scores indicate higher levels of treatment satisfaction for DTSQs items 1, 4 -8. For items 2 and 3 a higher score indicates a higher patient perceived experience of high blood sugars and low blood sugars, respectively. Thus, lower scores indicate a perception of blood glucose levels being "none of the time" unacceptably high (item 2) or low (item 3). The domain score of total treatment satisfaction (total treatment satisfaction score) was computed by adding the six items scores 1, 4-8. The score ranges 0-36. A higher treatment satisfaction score indicates a higher level of treatment satisfaction. Results are based on the data from the in-trial observation period.
Time Frame: Week 0, week 104
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Oral Semaglutide Flex- Sustainability
Number analyzed (Participants) | 180
Score on a scale
  1) Satisfaction with treatment | 1.19 (1.61)
  2) Feeling of unacceptably high blood sugars | -1.46 (2.44)
  3) Feeling of unacceptably low blood sugars | -0.14 (2.09)
  4) Convenience of treatment: number analyzed (Participants) | 179
  4) Convenience of treatment | 0.88 (1.52)
  5) Flexibility of current treatment | 0.86 (1.56)
  6) Satisfaction with understanding of diabetes: number analyzed (Participants) | 179
  6) Satisfaction with understanding of diabetes | 0.84 (1.50)
  7) Recommending treatment to others | 0.94 (1.58)
  8) Satisfaction to continue with present treatment | 1.11 (1.62)
  Total treatment satisfaction score | 5.81 (7.11)

ADVERSE EVENTS:
Time Frame: Week 0 to week 109. Results are based on the safety analysis set (SAS), which comprised all randomised participants who received at least one dose of trial product.
Description: Serious adverse events and other AEs were based on the on-treatment observation period, i.e., the time period when a participant was on treatment with trial product, including any period after initiation of rescue medication. All-cause mortality were based on the in-trial observation period, i.e., the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product.
Arm/Group | Oral Semaglutide Flex- Main Phase | Sitagliptin 100 mg- Main Phase | Oral Semaglutide Flex- Sustainability | Oral Semaglutide Flex- Switch | Sitagliptin 100 mg- Switch
All-Cause Mortality (participants affected / at risk) | 0/253 | 2/250 | 0/253 | 0/100 | 0/97
Serious Adverse Events (participants affected / at risk) | 24/253 | 24/250 | 36/253 | 9/100 | 7/97
Other Adverse Events (participants affected / at risk) | 126/253 | 70/250 | 148/253 | 46/100 | 27/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide Flex- Main Phase (N=253) | Sitagliptin 100 mg- Main Phase (N=250) | Oral Semaglutide Flex- Sustainability (N=253) | Oral Semaglutide Flex- Switch (N=100) | Sitagliptin 100 mg- Switch (N=97)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bladder prolapse (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Catheterisation cardiac (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Coronary artery insufficiency (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Intestinal mass (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Cataract operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gastric bypass (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Macular fibrosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Otitis media chronic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otosclerosis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian endometrioid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pharyngeal polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shoulder operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Semaglutide Flex- Main Phase (N=253) | Sitagliptin 100 mg- Main Phase (N=250) | Oral Semaglutide Flex- Sustainability (N=253) | Oral Semaglutide Flex- Switch (N=100) | Sitagliptin 100 mg- Switch (N=97)
Abdominal pain upper (Gastrointestinal disorders) | 16 (17) | 3 (3) | 20 (27) | 6 (6) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 22 (25) | 8 (11) | 29 (39) | 10 (11) | 3 (5)
Dyspepsia (Gastrointestinal disorders) | 13 (13) | 2 (4) | 18 (23) | 4 (4) | 2 (2)
Headache (Nervous system disorders) | 25 (33) | 15 (15) | 29 (47) | 4 (4) | 3 (3)
Nasopharyngitis (Infections and infestations) | 26 (30) | 13 (15) | 34 (58) | 7 (8) | 10 (11)
Nausea (Gastrointestinal disorders) | 53 (83) | 6 (8) | 58 (113) | 17 (19) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 15 (16) | 18 (33) | 1 (2) | 4 (5)
Vomiting (Gastrointestinal disorders) | 14 (21) | 2 (2) | 18 (39) | 7 (8) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (12) | 8 (9) | 17 (34) | 3 (5) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (14) | 11 (14) | 17 (34) | 3 (3) | 5 (5)
Constipation (Gastrointestinal disorders) | 7 (9) | 7 (8) | 11 (17) | 5 (5) | 1 (1)
Gastroenteritis (Infections and infestations) | 9 (9) | 1 (1) | 13 (19) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 10 (11) | 6 (8) | 15 (23) | 6 (6) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT02849080/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT02849080/SAP_001.pdf